CLINICAL TRIAL: NCT00552227
Title: The Effect of Protein Kinase C (PKC) β Specific Inhibitor on Oxidant Stress in Patient With Type 2 Diabetes Mellitus
Brief Title: Isoprostane/FMD Study The Effect of Protein Kinase C (PKC) β Specific Inhibitor LY333531 on Oxidant Stress in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6038; B7A-MC-MBCZ
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ruboxistaurin
- 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ruboxistaurin — oral 32 mg daily
  Other Names: LY333531
  Arms: 1
Other: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether ruboxistaurin can reduce blood vessel inflammation associated with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus
2. ≥35 years of age
3. Fasting low-density lipoprotein (LDL) cholesterol <160 mg/dL, triglycerides (TG) <400 mg/dL
4. Sitting systolic blood pressure <160 mm Hg and sitting diastolic blood pressure <90 mm Hg as determined by the mean of three separate measurements.
5. Hemoglobin A1c (HbA1c) ≥7% and ≤11%.

   Exclusion Criteria:
6. A serum creatinine >2.0 mg/dL or who have received a renal transplant or are currently being treated with dialysis.
7. Alanine aminotransaminase (ALT), alkaline phosphatase (ALP), or total bilirubin (TB) greater than two times the upper limit of normal
8. Current use of aspirin, nitroglycerin or long-acting nitrates or potential need for use of aspirin, nitroglycerin or long-acting nitrates to treat documented cerebrovascular or coronary artery disease during the study.
9. Use of tobacco products (for example, cigarettes, cigars, pipes, and snuff) within the 6 months prior to Visit 1.
10. Requirement for treatment with very potent inhibitors of cytochrome P450 3A4 or inhibitors of cytochrome P450 2D6.
11. Requirement for treatment with inducers of cytochrome P450 3A4.
12. Active infection/inflammation as determined by body temperature >38°C OR current use of systemic antibacterial, antifungal, or antiviral medication OR active chronic inflammation (for example, lupus, rheumatoid arthritis, multiple sclerosis).
13. Abdominal, thoracic, vascular, or cranial surgery that is determined to be of major significance by the investigator within 3 months prior to Visit 1.
14. Current suspicion of carcinoma or treatment for cancer within 6 months prior to Visit 1 or anticipated treatment for cancer during the course of the study, with the exception of superficial lesions such as basal cell carcinoma and squamous cell carcinoma of the skin.
15. Patients who have taken any non-steroidal anti-inflammatory agents (including aspirin and cyclooxygenase-2 inhibitors) or vitamins within 14 days of entry (Visit 1).
16. Patients who have previously completed or withdrawn from this study or any other study investigating LY333531 (unless the patient is being re-screened 14 days or more after discontinuing the use of vitamins or non-steroidal anti-inflammatory agents.
17. Directly affiliated with the conduct of this study, or are immediate family of someone directly affiliated with the conduct of this study (that is, Lilly employees, investigators, site personnel, or their immediate families). Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
18. Treatment with an investigational drug within the last 30 days at the time of study entry.
19. Females of child-bearing potential (not surgically sterilized and between menarche and <5 years post menopause) who test positive for pregnancy at the time of enrollment based on a serum pregnancy test or who intend to become pregnant during the study.
20. Females of child-bearing potential who do not agree to use a reliable method of birth control (for example, use of oral contraceptives or Norplant®; a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices]; partner with vasectomy; or abstinence) during the study.
21. A female who is breast-feeding.
22. Any other findings, in the opinion of the investigator, that would preclude the patient's participation in the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-09; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measure is the ratio of urinary isoprostane to creatinine as measured by gas chromatography/mass spectrometry (GC/MS) in the two consecutive 12-hour urine samples obtained prior to both Visit 2 (baseline) and Visit 3 (endpoint). | 6 weeks

SECONDARY OUTCOMES:
Increase in brachial artery diameter induced by reactive hyperemia as measured by ultrasound (flow-mediated dilatation) at Visits 2 and 3. | 6 weeks
The ratio of urinary albumin to creatinine | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muredach Reilly, MD, Principal Investigator — University of Pennsylvania, Philadelphia
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 am to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com